CLINICAL TRIAL: NCT01571531
Title: European Multicentre Study of Human SCI
Brief Title: European Multicentre Study of Human Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK-03/2004 / PB_2016-00293
Record Dates: First submitted 2012-04-02; First posted 2012-04-05 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Today there is accumulating evidence from animal experiments that regeneration can be induced after a spinal cord injury (SCI). Consequently in the near future, new therapeutic approaches to induce some regeneration will be included in the treatment of patients with SCI. The aim of this proposal is to provide the required clinical basis for the implementation of novel interventional therapies. The establishment of combined clinical, functional and neurophysiological measures for a qualitative and quantitative assessment of spinal cord function in patients with SCI at different stages during rehabilitation represents a basic requirement to monitor any significant effect of a new treatment. Therefore, several European Paraplegic Centres involved in the rehabilitation of acute traumatic SCI patients build up a close collaboration for standardised assessment. The aim is to get knowledge about the natural recovery after spinal cord lesion in a larger population of patients in the sense of a historical control group and to bring new standardised assessment tools to the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Single event traumatic or ischemic para- or tetraplegia
* First EMSCI assessment possible within the first 6 weeks after incidence
* Patient capable and willing of giving written informed consent

Exclusion Criteria:

* Nontraumatic para- or tetraplegia (i.e. discusprolaps, tumor, AV-malformation, myelitis) excl. single event ischemic incidences
* Pre-known dementia or severe reduction of intelligence, leading to reduced capabilities of cooperation or giving consent
* Peripheral nerve lesions above the level of lesion (i.e. plexus brachialis impairment)
* Pre-known polyneuropathy
* Severe craniocerebral injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2004-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Independence Measure (SCIM) | Change in course from 2 weeks at 48 weeks
  Score from 0 to 100 points; the higher the score, the higher the independence of the patient
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI score) | Change in course from 2 weeks at 48 weeks
  Score from 0 to 112; the higher the score, the better the neurological status of the patient
Walking Index for Spinal Cord Injury (WISCI) | Change in course from 2 weeks at 48 weeks
  Score from 0 to 20; the higher the score, the better the walking ability of the patient
10 Meter Walk Test (10mWT) | Change in course from 2 weeks at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Armin Curt, Prof., MD, Principal Investigator — University of Zurich; Martin Schubert, MD, Study Director — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Pavese C, Scivoletto G, Puci M, Rupp R, Schubert M, Rohrich F, Waldmann J, Weidner N, Kalke YB, Abel R, Maier D, Kriz J, Chhabra HS, Rehahn K, Montomoli C, Curt A, Jutzeler CR. The Relationship Between Age and Recovery After Spinal Cord Injury: A Longitudinal Cohort Study. Neurology. 2026 Jan 27;106(2):e214516. doi: 10.1212/WNL.0000000000214516. Epub 2025 Dec 23. PMID 41428979
- [Derived] Sliwinski C, Heutehaus L, Taberner FJ, Weiss L, Kampanis V, Tolou-Dabbaghian B, Cheng X, Motsch M, Heppenstall PA, Kuner R, Franz S, Lechner SG, Weidner N, Puttagunta R. Contribution of mechanoreceptors to spinal cord injury-induced mechanical allodynia. Pain. 2024 Jun 1;165(6):1336-1347. doi: 10.1097/j.pain.0000000000003139. Epub 2023 Dec 27. PMID 38739766
- [Derived] Pavese C, Scivoletto G, Puci MV, Abel R, Curt A, Maier D, Rupp R, Schubert M, Weidner N, Montomoli C, Kessler TM. Prediction of bowel management independence after ischemic spinal cord injury. Eur J Phys Rehabil Med. 2022 Oct;58(5):709-714. doi: 10.23736/S1973-9087.22.07366-X. Epub 2022 Jun 6. PMID 35666490
- [Derived] Franz S, Rust L, Heutehaus L, Rupp R, Schuld C, Weidner N. Impact of Heterotopic Ossification on Functional Recovery in Acute Spinal Cord Injury. Front Cell Neurosci. 2022 Feb 9;16:842090. doi: 10.3389/fncel.2022.842090. eCollection 2022. PMID 35221928
- [Derived] Buri M, Curt A, Steeves J, Hothorn T. Baseline-adjusted proportional odds models for the quantification of treatment effects in trials with ordinal sum score outcomes. BMC Med Res Methodol. 2020 May 6;20(1):104. doi: 10.1186/s12874-020-00984-2. PMID 32375705
- See also: Related Info — http://www.emsci.org